CLINICAL TRIAL: NCT01998867
Title: Identification of Fasting Biomarkers That Predict Responses to the Oral Glucose Tolerance Test (OGTT) and Mixed Meal Tolerance Test (MMTT)
Brief Title: Fasting Predictors of OGTT and MMTT Response
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Health Diagnostic Laboratory, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: R2013-1003
Record Dates: First submitted 2013-11-25; First posted 2013-12-02 (Estimated); Last update posted 2015-02-13 (Estimated); Status verified 2015-02

CONDITIONS: Prediabetes; Hypertension; Obesity; Cardiovascular Disease
MeSH Terms: conditions — Prediabetic State; Hypertension; Obesity; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood and serum
Oversight: Data Monitoring Committee: No

SUMMARY:
1. To develop a database containing matched information from dynamic tests of postprandial glycemic control (OGTT or MMTT), results of a broad panel of fasting biomarkers, and clinical information related to diabetes risk obtain through subject interview.
2. To use the database to identify fasting biomarkers and associated algorithms to best predict parameters derived from dynamic tests (OGTT or MMTT) such as Insulin Glucose Tolerance (IGT), impaired first phase insulin response, etc., controlling for clinical information such as current medication use.

ELIGIBILITY:
Inclusion Criteria:

* Weight >95

Exclusion Criteria:

* Prior diagnosis of Diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Representative of the ethnic population of Richmond, VA
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2013-08; Primary Completion 2018-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Identify fasting biomarkers and associated algorithms to predict parameters | Baseline
  To assess relations between baseline factors and patterns of change over time due to feeding treatments.

CONTACTS AND LOCATIONS:
Overall Officials: Szilard Voros, MD, Principal Investigator — Health Diagnostic Laboratory, Inc.
Locations (1):
- Health Diagnostic Laboratory, Inc., Richmond, Virginia, United States

REFERENCES:
- [Background] Go AS, Mozaffarian D, Roger VL, Benjamin EJ, Berry JD, Borden WB, Bravata DM, Dai S, Ford ES, Fox CS, Franco S, Fullerton HJ, Gillespie C, Hailpern SM, Heit JA, Howard VJ, Huffman MD, Kissela BM, Kittner SJ, Lackland DT, Lichtman JH, Lisabeth LD, Magid D, Marcus GM, Marelli A, Matchar DB, McGuire DK, Mohler ER, Moy CS, Mussolino ME, Nichol G, Paynter NP, Schreiner PJ, Sorlie PD, Stein J, Turan TN, Virani SS, Wong ND, Woo D, Turner MB; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Executive summary: heart disease and stroke statistics--2013 update: a report from the American Heart Association. Circulation. 2013 Jan 1;127(1):143-52. doi: 10.1161/CIR.0b013e318282ab8f. No abstract available. PMID 23283859
- [Background] Roger VL, Go AS, Lloyd-Jones DM, Benjamin EJ, Berry JD, Borden WB, Bravata DM, Dai S, Ford ES, Fox CS, Fullerton HJ, Gillespie C, Hailpern SM, Heit JA, Howard VJ, Kissela BM, Kittner SJ, Lackland DT, Lichtman JH, Lisabeth LD, Makuc DM, Marcus GM, Marelli A, Matchar DB, Moy CS, Mozaffarian D, Mussolino ME, Nichol G, Paynter NP, Soliman EZ, Sorlie PD, Sotoodehnia N, Turan TN, Virani SS, Wong ND, Woo D, Turner MB; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Executive summary: heart disease and stroke statistics--2012 update: a report from the American Heart Association. Circulation. 2012 Jan 3;125(1):188-97. doi: 10.1161/CIR.0b013e3182456d46. No abstract available. PMID 22215894
- [Background] DeFronzo RA, Abdul-Ghani M. Type 2 diabetes can be prevented with early pharmacological intervention. Diabetes Care. 2011 May;34 Suppl 2(Suppl 2):S202-9. doi: 10.2337/dc11-s221. PMID 21525456
- [Background] Nathan DM, Davidson MB, DeFronzo RA, Heine RJ, Henry RR, Pratley R, Zinman B; American Diabetes Association. Impaired fasting glucose and impaired glucose tolerance: implications for care. Diabetes Care. 2007 Mar;30(3):753-9. doi: 10.2337/dc07-9920. No abstract available. PMID 17327355